CLINICAL TRIAL: NCT06750588
Title: Phase 1, Open Label Study to Evaluate Safety and Tolerability of NTR-101 in Patients With Acute Alcohol-Associated Hepatitis
Brief Title: Safety and Tolerability of NTR-101 in Patients With Acute Alcohol-Associated Hepatitis
Acronym: PhoenixAH
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nterica Bio inc (Industry)
Collaborators: Southern California Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NtericaAH-001
Record Dates: First submitted 2024-11-29; First posted 2024-12-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Alcohol-Associated Hepatitis
Keywords: bacteriophages; alcohol-associated hepatitis; NTR-101; bacteriophage therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Active Comparator): Dose 1
  Interventions: Drug: bacteriophage preparation
- Cohort 2 (Active Comparator): Dose 2
  Interventions: Drug: Bacteriophage preparation
- Cohort 3 (Active Comparator): Dose 3
  Interventions: Drug: bacteriophage preparation
- Cohort 4 (Active Comparator): Dose 4
  Interventions: Drug: bacteriophage preparation

INTERVENTIONS:
Drug: bacteriophage preparation — NTR-101 will be given orally to participants once daily for 7 days
  Arms: Cohort 1
Drug: Bacteriophage preparation — NTR-101 will be given orally to participants once daily for 7 days
  Arms: Cohort 2
Drug: bacteriophage preparation — NTR-101 will be given orally to participants twice daily for 7 days
  Arms: Cohort 3
Drug: bacteriophage preparation — NTR-101 will be given orally to participants three times daily for 7 days
  Arms: Cohort 4

SUMMARY:
The goal of this clinical trial is to learn about the safety and tolerability of NTR-101 in adult participants suffering from acute alcohol-associated hepatitis (AH).

The drug is intended for use in the treatment of AH where the presence of specific strains of E. faecalis play a contributing role.

The main questions it aims to answer are:

Are multiple doses of NTR-101 in participants with acute AH safe and well tolerated? What medical problems do participants have when taking NTR-101? Researchers will administer the drug and monitor participants in an inpatient center.

Participants will:

Be administered multiple ascending dose frequencies of NTR-101 every day for 7 days.

Stay in the clinic for 9 days (7 days of treatment) and present to clinic once every week for checkups and tests for 35 days.

Keep a diary of their symptoms until the checkups and tests are completed.

DETAILED DESCRIPTION:
Alcohol-associated hepatitis (AH) is a severe inflammatory liver disease that can progress to liver failure, with high morbidity and mortality rates. Emerging studies indicate a significant role of gut-derived pathogens, particularly Enterococcus faecalis (E faecalis), in exacerbating liver damage through bacterial translocation and the release of toxins.

Cytolysin-positive E. faecalis strains exhibit high virulence and resistance to standard antibiotics.

NTR-101 is a product developed for oral delivery and composed of natural bacteriophages that specifically target cytolysin-positive E. faecalis.

The targeted activity of NTR-101 against E. faecalis in AH patients has the potential to address the underlying bacterial trigger, offering a novel approach to mitigate liver inflammation and reduce disease progression. For patients who do not respond to traditional treatments like corticosteroids or experience reduced antibiotic therapy efficacy, NTR-101 represents a novel, targeted approach that leverages bacteriophages' specificity for bacterial strains in this target population, offering a potential alternative or complement to traditional antibiotics.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnostic definition of acute alcohol-associated hepatitis based on well established standard disease markers
* Able to provide written informed consent (either from patient or patient's legally authorized representative)
* Male and female patients aged ≥18 years and ≤ 70 years of age
* BMI ≥ 20 to ≤ 40 kg/m2
* Enterococcus faecalis testing
* Susceptibility to NTR-101
* Women of child-bearing potential and male patients must agree to use a medically acceptable method of contraception/ birth control throughout the study duration.

Key Exclusion Criteria:

* Participants considered at high risk for alcohol withdrawal according to the clinical institute withdrawal assessment (CIWA-Ar) protocol
* Participants taking systemic corticosteroids for a specified duration
* Platelet count below specified ranges
* INR and Serum creatinine levels above specified ranges
* Active bacterial or viral infections
* Other or concomitant cause(s) of liver disease as a result of other conditions
* Co-infection with HIV
* Positive urine drug screen
* Any significant systemic or major illness other than liver disease that, in the opinion of the investigator, would preclude the patient from participating in and completing the study or might complicated or exacerbated by the proposed treatments or might confound assessment of investigational product
* If female, known pregnancy, or has a positive serum pregnancy test, or lactating/ breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | AEs will be recorded daily for 7 days, then weekly on days 14, 21, 28 and 35
  The number of adverse events (AEs) will be recorded.
Changes in liver function will be evaluated | Assessments will be recorded daily for 7 days, then weekly on days 14, 21, 28 and 35
  ALT (alanine transaminase) and AST (aspartate aminotransferase) enzymes will be evaluated

SECONDARY OUTCOMES:
Preliminary assessment of NTR-101 efficacy and viability | Stool samples will be collected daily for 7 days, then weekly on days 14, 21, 28 and 35 to evaluate the presence of the target pathogen and NTR-101 viability
  Assessment of relative abundance of target pathogen and NTR-101 viability after oral administration

OTHER OUTCOMES:
Evaluation of the effect of NTR-101 on various disease severity markers | Samples for disease severity markers be collected daily for 7 days, then weekly on days 14, 21, 28 and 35
  changes from baseline in disease severity markers like Serum bilirubin, Serum sodium, Serum creatinine
Susceptibility of recovered target bacteria to NTR-101 post-treatment | Samples will be collected daily for 7 days, then weekly on days 14, 21, 28 and 35
  Stool samples will be collected for bacteria culture and assess for susceptibility to NTR-101

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hassanein, MD, Principal Investigator — Southern California Research Center, inc
Locations (1):
- Southern California Research Center, inc, Coronado, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
The study IPD may not be shared for three key reasons.
  1. The study is primarily designed to assess the safety and tolerability of a drug in a small group of participants, making the sample size too small to ensure participant anonymity. Revealing individual data could risk participant privacy, especially as the study is open label.
  2. This study is also aimed at collective sensitive information regarding pharmacokinetics, dosing levels, and early safety signals, which are critical to a sponsor's competitive advantage. Sharing this data prematurely could impact intellectual property or strategic positioning at this early stage of development.
  3. This study is not aimed to demonstrating efficacy but rather focus on basic safety and dose-ranging, making the data limited in broader scientific value compared to later-phase trials.

REFERENCES:
- [Background] Mendes BG, Duan Y, Schnabl B. Immune Response of an Oral Enterococcus faecalis Phage Cocktail in a Mouse Model of Ethanol-Induced Liver Disease. Viruses. 2022 Feb 27;14(3):490. doi: 10.3390/v14030490. PMID 35336897
- [Background] Duan Y, Llorente C, Lang S, Brandl K, Chu H, Jiang L, White RC, Clarke TH, Nguyen K, Torralba M, Shao Y, Liu J, Hernandez-Morales A, Lessor L, Rahman IR, Miyamoto Y, Ly M, Gao B, Sun W, Kiesel R, Hutmacher F, Lee S, Ventura-Cots M, Bosques-Padilla F, Verna EC, Abraldes JG, Brown RS Jr, Vargas V, Altamirano J, Caballeria J, Shawcross DL, Ho SB, Louvet A, Lucey MR, Mathurin P, Garcia-Tsao G, Bataller R, Tu XM, Eckmann L, van der Donk WA, Young R, Lawley TD, Starkel P, Pride D, Fouts DE, Schnabl B. Bacteriophage targeting of gut bacterium attenuates alcoholic liver disease. Nature. 2019 Nov;575(7783):505-511. doi: 10.1038/s41586-019-1742-x. Epub 2019 Nov 13. PMID 31723265